CLINICAL TRIAL: NCT07165522
Title: Adapting and Testing a Novel Method of Engagement in Research: Centering Autistic Perspectives in Behavioral Intervention Discussions
Brief Title: Centering Autistic Perspectives in Behavioral Intervention Discussions
Acronym: CAPBID SoE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, Matthew Lerner, Associate Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2507011294
Record Dates: First submitted 2025-08-21; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Autism
Keywords: Autism; Applied Behavior Analysis; ABA; Community Based Participatory Research; Transformative and Restorative Justice; Engagement
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Quantitative data analysts will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transformative and Restorative Engagement Circle (TREC) (Experimental)
  Interventions: Behavioral: Transformative and Restorative Engagement Circle (TREC)
- Stakeholder Engagement in quEstion Development and prioritization (SEED) (Active Comparator)
  Interventions: Behavioral: Stakeholder Engagement in quEstion Development and prioritization (SEED)

INTERVENTIONS:
Behavioral: Transformative and Restorative Engagement Circle (TREC) — TREC will be co-developed in Phase 1, to focus on ensuring the presence of at least 3 key components: 1) a listening phase (focused on unconditionally hearing the experiences of autistic participants), 2) an acknowledgement phase (in which the experiences, including but not limited to harms and trauma, of autistic participants will be expressly addressed and acknowledged), 3) a negotiation/priority-setting phase, in which participants will collaboratively identify goals for future CER.
  Arms: Transformative and Restorative Engagement Circle (TREC)
Behavioral: Stakeholder Engagement in quEstion Development and prioritization (SEED) — The SEED Method is a PCORI-supported multilevel stakeholder engagement model, using a participatory framework to develop stakeholder priorities. The core premise of SEED is creating a level playing field for stakeholders, wherein participants learn how to collaboratively identify their own community's priorities, and then refine them together. It involves convening participatory Topic Groups of stakeholders, assembled based on their experience and knowledge of the area of focus (in this case, autism and ABA). It also involves additional consultative stakeholder participants to fill in key gaps in representation; this element may or may not be present in thi SEED iteration, based on the CAC-led adaptation. SEED participants convene over a period of time (adapted to the needs of the specific group, and will be matched to the length of TREC here) to conceptualize (i.e., learn how to build a conceptual model and conduct exercises to do so), generate questions (i.e., review the conceptual m
  Arms: Stakeholder Engagement in quEstion Development and prioritization (SEED)

SUMMARY:
The Centering Autistic Perspectives for Behavioral Interventions Discussions (CAPBID) PCORI Science of Engagement Award will examine different community engagement approaches for bringing together autistic people, Applied Behavioral Analysis (ABA) providers, and other members of the autism community to advance a shared equitable dialogue around research priorities for ABA-related research. One of these approaches will be based on existing transformative and restorative justice methods and frameworks. This project also utilizes a community-driven participatory research approach that will center autistic leadership in all aspects of the project.

The investigators hope that this research will pave the way for creating spaces where autistic people are heard in their experiences and can collaborate effectively with open-minded ABA providers about how to advance the next generation of care and research in the field. More broadly, the investigators aim to create engagement approaches that may be used to have conversations around critical and difficult issues faced by the autistic and autism communities, as well as other marginalized communities.

DETAILED DESCRIPTION:
Ensuring systematically marginalized populations have access to clinical care that is accessible and meaningful is a vital public health issue. However, many such communities have concerns about available supports and/or lack trust in researchers that study them, precluding advancement of the very comparative clinical effectiveness research (CER) that could address these needs. It is presently unknown what engagement approaches are best suited to bring patients and other stakeholders together to develop shared CER priorities. While frameworks exist for such engagement, no rigorous, comparative research on consequent methods yet exists.

An urgent instance of this gap is the relationship between the autistic community and Applied Behavior Analysis (ABA)-based intervention, which is both viewed as uniformly beneficial by practitioners and enshrined in law by policymakers yet is increasingly denounced and viewed as harmful by autistic adults. This yields a growing chasm between the care that is most widely available to this population, and the willingness of autistic people and their families to engage with it - begging the question of what engagement approach can begin to bridge this rift.

One common approach to bringing stakeholders together to advance CER is to engage them in equitable shared decision-making processes. However, some evidence suggests there may be a unique value to centering marginalized perspectives to more effectively promote equity of engagement and prioritization of CER goals acceptable to the full range of stakeholders. Transformative and Restorative Justice practices offer methods for engagement that offer such centering, particularly around circumstances where some have experienced harm. Thus, a comparison of such approaches, applied to the autism and ABA debate, offers a rich opportunity to both address a pressing needed in this specific community, and identify effective methods for CER engagement in marginalized communities more broadly.

Study Aims:

To develop a Transformative and Restorative Engagement Circle (TREC) approach for centering autistic people in ABA-related CER priority setting.

To compare TREC and SEED approaches on their impacts on engagement with autistic adults & autism stakeholders.

Utilize a partially-masked randomized control trial (RCT) to compare the TREC approach to an established equity-focused approach called Stakeholder Engagement in quEstion Development and prioritization (SEED) approach.

Evaluate the impact on measures of patient and stakeholder buy-in, agency, collective goal setting, and ongoing engagement before, during, and after participating in either the TREC or SEED approaches.

Understand barriers and facilitators for successful engagement.

To compare TREC and SEED approaches in terms of acceptability and importance of identified CER priorities within the broader autistic patient and autism stakeholder communities.

The investigators will field a national survey across the autism community, to assess the relative acceptability of TREC- vs. SEED-derived CER priorities.

Study Description:

The investigators will conduct a three-phase mixed methods study to develop and test the proposed TREC and SEED engagement approaches (EA) and examine the acceptability and importance of the ABA-related CER priorities they produce.

First, investigators will co-develop the TREC EA utilizing participatory research methods in partnership between the CAPBID Leadership Team, autistic Community Advisory Council (CAC), and partnered Transformative and Restorative Justice facilitators. This co-development process will also yield a process by which procedural elements of TREC and SEED will be matched, and quantitative engagement measures will be co-adapted for the autistic community. This phase will take six months.

Second, investigators will conduct a mixed-method embedded randomized controlled trial (RCT) comparing two engagement methods, TREC and SEED. The key manipulation is that TREC centers autistic voices as an example of a marginalized patient population, whereas SEED aims to engage all stakeholders equally. 200 adult participants (100 autistic, 100 other stakeholders, including at least 40 ABA providers, 40 caregivers, and 20 policymakers) will be recruited over 1.5 years from team and partner networks, online fora, conferences, and other spaces representative of target groups. Stratified randomized based on stakeholder group and perspective on ABA appropriateness for autism will be used to assign participants to TREC or SEED. Participants will complete quantitative measures of (primary outcomes) accessibility, buy-in, trust, and collective goal-setting immediately before, at midpoint, and immediately following engagement activities; engagement quality will be measured at midpoint and endpoint. Both TREC and SEED will conclude with prioritization of ABA-related CER goals. (Secondary outcome) Willingness to engage in further ABA-related CER will be assessed at endpoint, 1-week, and 1-month follow-up. A subset will additionally complete qualitative interviews regarding barriers and facilitators to engagement, which will be analyzed thematically.

Finally, investigators will distill ABA-related CER priorities from TREC and SEED, which will then be fielded in a national American sample (n=500 adults; at least 100 autistic, 100 ABA provider, 100 caregiver, 100 researchers, 100 other stakeholders) recruited through online networks and community contacts to identify (primary outcome) differential acceptability of TREC- and SEED-derived priorities. This will take place over 6 months.

This study builds on the leadership of the Centering Autistic Perspectives in Behavioral Intervention Discussions (CAPBID) Leadership Team, a multistakeholder group of autistic people, researchers, scholars, ABA providers, and advocates working to center autistic perspectives in public discussions pertaining to behavioral interventions used in autism supports by directly acknowledging the lived experience of autistic people. The CAPBID team has been working together for more than 3 years to identify better ways to engage autistic people and autism stakeholders to advance more humane, person-centered care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 18
2. Individuals who have had experience with Applied Behavior Analysis (ABA) at any time in their lives who is:

   1. An Autistic individual who experienced Applied Behavior Analysis or
   2. A practitioner who currently or previously was involved in the delivery of Applied Behavior Analysis
3. Able to communicate fluently in English
4. Individuals who do not report the endpoint values on the AAPS:

   1. ABA should never be used for autistic people
   2. ABA is the only evidence-based intervention for autism

Exclusion Criteria:

1. Under the age of 18,
2. Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Brief Engagement Poll | Up to one day after the start of the intervention (engagement approach) delivery and up to 24 hours after completion of the intervention (engagement approach) delivery
  3-item poll indicating perceived quality ("ability to engage you as a member of our team in the meeting"), value ("Was today's meeting a good use of your time"), and contribution ("To what extent did you contribute to project-related processes") to the process, developed for autistic research partnerships by AASET
ABX Stakeholder Toolkit | At baseline, up to one day after the start of the intervention (engagement approach) delivery and up to 24 hours after the completion of the intervention (engagement approach) delivery
  Likert-type measure, with items including, "The study values the differences of contributing stakeholders," "I feel the study team has a clear understanding of stakeholders' expertise, strengths, and roles," "study stakeholders engage in open communication and demonstrate a willingness to listen to others," "My fellow stakeholder participants respect what I have to say, even when they do not agree with me." (post-engagement trust) "Participating in these activities has helped me better understand research on [this topic]," (sense of agency) "Individuals whose lives are most impacted by [this topic] are well represented," "I have decision-making authority and believe I contribute meaningfully to relevant outcomes and objectives for the study," "I feel that I have been compensated appropriately for my time and expertise as a stakeholder," "I have learned a lot from participating in these activities," "I feel I could explain the ABX study to others." (sense of buy-in)
Genetic Alliance Engagement Assessment Tool | At baseline, up to one day after the start of the intervention (engagement approach) delivery and up to 24 hours after the completion of the intervention (engagement approach) delivery
  Quantitative engagement metrics, including the degree to which "stakeholders report satisfaction in involvement in the research process and feel adequately informed about the project activities and results," and "Stakeholders report that the research is valuable to them and that they have contributed to setting and revising project priorities." as well as self-report items such as "A sense of partnership among team members and investigators has been established," "All team members are given equal opportunity to provide input," "Input from team members is incorporated into the decision-making process," and "There is clear communication about how input from team members is incorporated into decisions."

SECONDARY OUTCOMES:
ABA Willingness Tool | Up to 24 hours after completion of the intervention (engagement approach) delivery, up to 1-week after completion of the intervention, and up to 1-month after completion of the intervention.
  Likert-type measure regarding the willingness of participants to engage in further discussions regarding ABA-related CER. To be adapted with the CAC
AAPS | During screening for study enrollment and up to 1 week after completion of the intervention (engagement approach) delivery.
  1-item bipolar expanded -type self-report measure, indicating degree of pro- or anti-ABA positionality among participants. Scale endpoints will approximate, "I believe ABA should never be used with autistic people" and "All critiques of ABA are misguided, and ABA represents a uniformly useful evidence-based practice for autistic people."
AASPIRE CBPR Check In | At baseline, up to one day after the start of the intervention (engagement approach) delivery and up to 24 hours after the completion of the intervention (engagement approach) delivery
  A Likert-type measure, with items including "I feel I have the chance to say (or type) what I want to say during team meetings," "I feel like my comments are taken seriously," "I feel my opinions are valued" (sense of buy-in), and "this project is important," "I feel like this team works well together," "I find working on this project to be rewarding," "I am glad I am part of this team," "I am proud of the work we have done so far on this project" (post-engagement trust), all to be adapted with the CAC.
TREC and SEED Fidelity Tools | Up to 24 hours after each day of intervention (engagement approach)delivery.
  The Community Advisory Council-led process will yield co-development of a self-reported fidelity tool, to be completed by TREC Facilitators after each day. This tool will be used to assess the degree to which the groups adhered to the EA processes developed by the group
Qualitative Interviews | Up to three weeks after the completion of the intervention (engagement approach) delivery.
  Interviews up to 60 minutes. Semi-structured interview guide to be co-developed with the Community Advisory Council. Participant experience of EA, Barriers & facilitators to Engagement, Willingness to engage further regarding ABA-related CER

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Lerner, PhD, Principal Investigator — Drexel University; Dena L Gassner, PhD, Principal Investigator — Drexel University
Locations (1):
- AJ Drexel Autism Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Other investigators (e.g. Leadership Team) will obtain access to IPD as needed for trial completion.

REFERENCES:
- See also: PCORI Public Summary Page for this Project — https://www.pcori.org/research-results/2025/engagement-research-autistic-perspectives-behavioral-intervention